CLINICAL TRIAL: NCT01234714
Title: Liver Fat Quantification by Magnetic Resonance Imaging (MRI): A Novel Tool for Prediction of Postoperative Complications After Major Liver Resection?
Brief Title: Liver Fat Quantification by Magnetic Resonance Imaging (MRI) - Prediction of Postoperative Complications
Acronym: MRsteatosis
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: MRI_Steatosis_Outcomes
Record Dates: First submitted 2010-11-03; First posted 2010-11-04 (Estimated); Results first posted 2012-02-08 (Estimated); Last update posted 2012-02-08 (Estimated); Status verified 2012-02

CONDITIONS: Fatty Liver; Surgery
Keywords: Fatty Liver; Liver; Magnetic Resonance Imaging; Surgery
MeSH Terms: conditions — Fatty Liver | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Major liver resection: This single Cohort/Group will include all consecutive patients that received pre-operative Magnetic Resonant Imaging (MRI) and underwent major liver resection (>=3 segments).
  Interventions: Other: Non-invasive Magnetic Resonance Imaging (MRI); Procedure: Major liver resection

INTERVENTIONS:
Other: Non-invasive Magnetic Resonance Imaging (MRI) — Conventional pre-operative MRI
  Other Names: Magnetic Resonance Imaging
Procedure: Major liver resection — Hepatectomy of >= 3 liver segments
  Other Names: Hepatectomy = liver resection by open surgery.

SUMMARY:
The purpose of this study is to objectively quantify liver fat content (LFC) by Magnetic Resonant Imaging (MRI) prior to major liver surgery, and to investigate its association with post-operative complications.

DETAILED DESCRIPTION:
Lack of agreement exists among expert pathologists in the standard histological assessment of hepatic steatosis on biopsy. The impact of different grades of steatosis on postoperative complications after major liver resection remains controversial.

ELIGIBILITY:
Inclusion Criteria:

* Major liver resection (>= 3 resected segments).
* Patients that received a pre-operative Magnetic Resonance Imaging (MRI).
* Patient over 18 years of age

Exclusion Criteria:

* Patients that underwent liver surgery but < 3 segments were resected (e.g. wedge liver resection).
* Patient that did not receive a pre-operative MRI
* Patient age less than 18 years of age.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinics
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2010-10; Primary Completion 2010-12 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dimitri A Raptis, MD, MSc, Principal Investigator — University Hospital Zurich, Department of Visceral and Transplant Surgery, Zurich, Switzerland
Locations (2):
- Switzerland (2):
  - University Hospital Zurich, Department of Interventional and Diagnostic Radiology, Zurich, Canton of Zurich
  - University Hospital Zurich, Department of Visceral and Transplant Surgery, Swiss Hepato-Pancreato-Biliary (HPB) Center, Zurich, Canton of Zurich

REFERENCES:
- [Background] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912
- [Result] Raptis DA, Fischer MA, Graf R, Nanz D, Weber A, Moritz W, Tian Y, Oberkofler CE, Clavien PA. MRI: the new reference standard in quantifying hepatic steatosis? Gut. 2012 Jan;61(1):117-27. doi: 10.1136/gutjnl-2011-300155. Epub 2011 Oct 13. PMID 21997548

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients that underwent liver surgery were recruited at the outpatient clinics.
Period: Overall Study
Arm/Group | Major Liver Resection
Started | 84
Completed | 84
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Major Liver Resection
Number analyzed (Participants) | 84
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 67
  >=65 years | 17
Age Continuous [Mean (Standard Deviation); unit: years] | 54 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 44
Region of Enrollment [Number; unit: participants]
  Switzerland | 84

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Liver Fat Content on MRI in Patients With Serious Post-operative Complications (Clavien-Dindo Grade ≥IV)
Description: Liver fat content, measured by MRI, uses the in-phase/out-of-phase imaging calculated in terms of fat signal fraction (FSF).
  The Clavien-Dindo Classification of Surgical Complications:
  Grade I: Any deviation from the normal postoperative course without the need for treatment. Grade II: Requiring pharmacological treatment with drugs. Grade III: Requiring surgical, endoscopic or radiological intervention. Grade IV: Life-threatening complication requiring IC/ICU-management. Grade V: Death of a patient
Time Frame: December 2010
Population: According to the Clavien-Dindo Classification of surgical complications: (please see) http://www.surgicalcomplication.info/
Measure: Median (Inter-Quartile Range); unit: Percentage of liver fat content
Groups:
- Clavien-Dindo Grade <IV Complications: Percentage of liver fat content on MRI in patients with Clavien-Dindo Grade <IV complications.
  No complications: Patients without any post-operative complications defined according to the Clavien-Dindo Classification.
  Grade 1: Any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic and radiological interventions. Allowed therapeutic regimens are: drugs as antiemetics, antipyretics, analgetics, diuretics and electrolytes and physiotherapy. This grade also includes wound infections opened at the bedside.
  Grade II: Requiring pharmacological treatment with drugs other than such allowed for grade I complications.
  Blood transfusions and total parenteral nutrition are also included.
  Grade III:Requiring surgical, endoscopic or radiological intervention
- Clavien-Dindo Grade ≥IV Complications: Percentage of liver fat content on MRI in patients with Clavien-Dindo Grade <IV complications.
  These are typically life-threatening complication (including CNS complications) requiring ICU management.
  Grade IVa: single organ dysfunction (including dialysis)
  Grade IVb: multi-organ dysfunction
Arm/Group | Clavien-Dindo Grade <IV Complications | Clavien-Dindo Grade ≥IV Complications
Number analyzed (Participants) | 75 | 9
Percentage of liver fat content | 1.3 [0.5 to 4.2] | 13.6 [7.6 to 18.9]

2. Secondary Outcome: Post-operative Alanine Transaminase (ALT) Levels
Description: Alanine Transaminase is commonly measured clinically as a part of a diagnostic evaluation of hepatocellular injury, to determine liver health.
Time Frame: December 2010
Population: According to the MRI liver fat content measurement.
Measure: Median (Inter-Quartile Range); unit: Units/liter
Groups:
- Patient Group With Liver Fat Content <10% on MRI; Patient Group With Liver Fat Content >10% on MRI: Pre-operative Magnetic Resonance Imaging (MRI) liver fat content measurement (in percentage).
Arm/Group | Patient Group With Liver Fat Content <10% on MRI | Patient Group With Liver Fat Content >10% on MRI
Number analyzed (Participants) | 69 | 15
Units/liter | 386 [262 to 486] | 1355 [1277 to 1894]

3. Secondary Outcome: Intra-operative Blood Loss
Description: Intra-operative blood loss was defined according to the total volume of blood loss from the beginning until the end of the operation.
Time Frame: December 2010
Population: According to MRI
Measure: Median (Inter-Quartile Range); unit: ml
Arm/Group | Patient Group With Liver Fat Content <10% on MRI | Patient Group With Liver Fat Content >10% on MRI
Number analyzed (Participants) | 69 | 15
ml | 300 [200 to 500] | 400 [300 to 600]

4. Secondary Outcome: Operative Time
Description: The operation duration was measured according to the total minutes from the beginning of the operation until the end.
Time Frame: December 2010
Population: According to MRI
Measure: Median (Inter-Quartile Range); unit: min
Arm/Group | Patient Group With Liver Fat Content <10% on MRI | Patient Group With Liver Fat Content >10% on MRI
Number analyzed (Participants) | 69 | 15
min | 323 [240 to 405] | 360 [300 to 420]

5. Secondary Outcome: Intensive Care Unit (ICU) Stay
Description: The Intensive Care Unit (ICU) stay was calculated according to the total number of days the patients were managed in the ICU. This included also multiple ICU admissions.
Time Frame: December 2010
Population: According to MRI
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Patient Group With Liver Fat Content <10% on MRI | Patient Group With Liver Fat Content >10% on MRI
Number analyzed (Participants) | 69 | 15
days | 1 [1 to 1] | 2 [1 to 13]

6. Secondary Outcome: Hospital Stay
Description: The patient hospital stay was calculated according to the total number of days the patient was hospitalized.
Time Frame: December 2010
Population: According to MRI
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Patient Group With Liver Fat Content <10% on MRI | Patient Group With Liver Fat Content >10% on MRI
Number analyzed (Participants) | 69 | 15
days | 12 [10 to 16] | 19 [14 to 31]

7. Secondary Outcome: Cost
Description: The total in-hospital costs were calculated for each patient in Euros.
Time Frame: December 2010
Population: According to MRI
Measure: Mean (Standard Deviation); unit: Euros
Arm/Group | Patient Group With Liver Fat Content <10% on MRI | Patient Group With Liver Fat Content >10% on MRI
Number analyzed (Participants) | 69 | 15
Euros | 30363 (12701) | 83329 (86120)

8. Secondary Outcome: Type of Post-operative Complications
Description: There are several different types of post-operative complications associated with liver surgery, such as liver failure, multi-organ failure, bleeding, bile leak, and sepsis.
Time Frame: December 2010
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Time from MRI to patient hospital discharge after major liver resection.
Description: Serious and/or other [non-serious] adverse events were not collected/assessed.
Arm/Group | Major Liver Resection
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes